CLINICAL TRIAL: NCT04239196
Title: Open Label Phase II Randomized Non-comparative Study of SC Tocilizumab Associated With IV Pulse Steroid Versus IV Pulse Steroid Alone for the Treatment of Acute Anterior Ischemic Optic Neuropathy Associated With Giant Cell Arteritis
Brief Title: Efficacy of Tocilizumab for the Treatment of Acute AION Related to GCA
Acronym: TOCIAION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Roche Chugai (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17-03; 2019-001145-40 (EudraCT Number)
Record Dates: First submitted 2019-11-19; First posted 2020-01-23 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Giant Cell Arteritis; Optic Ischaemic Neuropathy
MeSH Terms: conditions — Giant Cell Arteritis; Optic Neuropathy, Ischemic | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: optimal Simon two-stage design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tocilizumab and IV steroids combination (Experimental): Every patient will receive the reference treatment for GCA with ocular complication, i.e. high dose corticosteroid therapy (intravenous pulses of 7,5 to 15 mg/kg/day of methylprednisolone with an upper limit of 1000 mg/day for 3 days followed by oral prednisone at 1 mg/kg/day with progressive decrease as usually done) and aspirin 75 mg/day. The mean duration of this reference treatment is 18 months. Patients will receive in addition to the reference treatment four subcutaneous injections of tocilizumab 162 mg over one month (1 injection per week).
  Interventions: Drug: tocilizumab and IV steroids combination
- IV steroids combination alone (Other): Every patient will receive the reference treatment for GCA with ocular complication, i.e. high dose corticosteroid therapy (intravenous pulses of 7,5 to 15 mg/kg/day of methylprednisolone with an upper limit of 1000 mg/day for 3 days followed by oral prednisone at 1 mg/kg/day with progressive decrease as usually done) and aspirin 75 mg/day. The mean duration of this reference treatment is 18 months.
  Interventions: Other: IV steroids combination alone

INTERVENTIONS:
Drug: tocilizumab and IV steroids combination — Every patient will receive the reference treatment for GCA with ocular complication, i.e. high dose corticosteroid therapy (intravenous pulses of 7,5 to 15 mg/kg/day of methylprednisolone with an upper limit of 1000 mg/day for 3 days followed by oral prednisone at 1 mg/kg/day with progressive decrease as usually done) and aspirin 75 mg/day. The mean duration of this reference treatment is 18 months.
  Patients will receive in addition to the reference treatment four subcutaneous injections of tocilizumab 162 mg over one month (1 injection per week).
  Arms: tocilizumab and IV steroids combination
Other: IV steroids combination alone — Every patient will receive the reference treatment for GCA with ocular complication, i.e. high dose corticosteroid therapy (intravenous pulses of 7,5 to 15 mg/kg/day of methylprednisolone with an upper limit of 1000 mg/day for 3 days followed by oral prednisone at 1 mg/kg/day with progressive decrease as usually done) and aspirin 75 mg/day. The mean duration of this reference treatment is 18 months.
  Arms: IV steroids combination alone

SUMMARY:
AION is the main cause of blindness in patients with GCA. High dose steroid is the reference treatment of this condition, but medical unmet need remains. Subcutaneous tocilizumab, a targeted biotherapy, recently received marketing authorization for the treatment of GCA, but only demonstrated at yet that it can allow steroid dose sparing. The aim of this study is to assess the benefit of tocilizumab and IV steroids combination or IV steroids alone, in the treatment of AION due to GCA.

DETAILED DESCRIPTION:
Tocilizumab will be proposed to eligible patients as an emergency treatment, in addition to the standard high-dose steroid treatment. Each patient will receive the reference treatment, i.e. one pulse of high dose intravenous methylprednisolone per day during 3 days, followed by 1 mg/kg/day oral prednisone, and low dose aspirin. Depending on the randomization, each patient will receive the reference treatment only, or will received in addition to the reference treatment four subcutaneous injections of tocilizumab 162 mg over one month (1 injection per week), the first tocilizumab injection being delivered on the same day than the first steroid IV pulse. Study visits will take place at 4, 8 and 13 weeks. The primary endpoint will be the ocular improvement at W8, defined as an increase of at least two lines of visual acuity on the ETRS chart. For each patient, the duration of participation will by of 3 months. The study duration is expected to be 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 50 years or older
2. Social insurance
3. Diagnosis of AION, characterized by sudden and painless loss of vision, of less than one week, accompanied by pallid swelling of the optic disc
4. Sudden permanent visual loss due to AION, of less than one week
5. Diagnosis of GCA based on the 1st (age ≥ 50 years) and the 3rd (Diagnosis of AION) criteria and at least one among the following :

   * One unequivocal symptom among: New onset localized headache, scalp or temporal artery tenderness, otherwise unexplained mouth or jaw pain under mastication, or unequivocal symptoms of polymyalgia rheumatic (shoulder and/or hip girdle pain associated with inflammatory stiffness).
   * Elevated erythrocyte sedimentation rate (≥ 50 at 1 hour) or C-reactive protein (≥ 10 mg/l), otherwise unexplained
   * Abnormal artery biopsy Biopsy specimen with artery showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells.
   * Evidence of large or medium-size vessel vasculitis at ultrasound, magnetic resonance angiography, computed tomography angiography, or positron emission tomography-computed tomography.

Exclusion Criteria:

* Other ocular involvements related to GCA (central retinal artery occlusion, posterior ischemic optic neuropathy, transient ocular manifestations, occipital stroke), if not associated with AION
* Biological targeting therapy within 3 months preceding the study
* Evidence of active infection
* History of any malignant neoplasm except adequately treated basal or squamous cell carcinoma of the skin or solid tumors treated with curative therapy and disease-free for at least 5 years
* History of recurrent infections, diverticulitis or intestinal ulceration and ASAT/ALAT > 5 * upper limit of normal, according to the Summary of Product Characteristics of tocilizumab
* Contraindication to steroids and/or aspirin administrated in the treatment
* Breastfeeding women and women with childbearing potential without highly effective contraception.
* Pregnant or nursing (lactating) women confirmed by a positive βHCG laboratory test at the inclusion
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during study treatment and for 3 months after the last administration of tocilizumab.
* Cytopenia, as defined by platelet count < 100 × 109/L (100,000/mm3), hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L), absolute neutrophil count < 2.0 × 109/L (2000/mm3), absolute lymphocyte count < 0.5 × 109/L (500/mm3)
* Insufficient liver function (Child Pugh C )
* Insufficient kidney function, as defined by a serum creatinine of more than 3 mg/dL or creatinine clearance of 20 ml/min or less
* Patients with previously untreated tuberculosis, previously known TDM/radiographic evidence suggestive of active and/or sequellar tuberculosis
* HIV infected, hepatitis C infected, or a positive hepatitis B surface antigen if known before study inclusion
* Contraindication to and precaution in use of tocilizumab according to the summary product description
* Inability to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
ocular change | Week 8
  The primary endpoint will be the ocular change at Week 8. This change will be defined as the increase of at least two lines of visual acuity on the ETDRS chart.

SECONDARY OUTCOMES:
Decrease of vision | Week 8
  Stabilization of vision, as judged at Week 8 after treatment start, correspond to a lack of deterioration :
  * If the patient can see the light initially, no light perception at W8 will represent a deterioration
  * If the patient is able to count finger at any distance, but the visual acuity is less than 20/400 on the ETRS chart, a "off chart" visual acuity at W8 will represent a deterioration
  * If initial visual acuity is equal or more than 20/400, a loss of 2 lines or more on the ETDRS at Week 8 will represent deterioration
Occurrence of a visual improvement | Week 4 and Week 13
  Occurrence of a visual improvement defined as an increase of two lines or more of visual acuity on ETDRS chart, a clinically significant difference, at Week 4 and Week 13
Change in Mean Deviation | weeks 4, 8, and 13
  Change in Mean Deviation (MD) measured on an automatized Visual Field (SITA Standard Humphrey 24-2) at weeks 4, 8, and 13
Changes in angio-OCT | Week 0 and Week 4
  Changes in angio-OCT between baseline and Week 4 : superficial and deep vascular plexus will be examined to look for the decrease of ischemia in peripapillary and macular areas.
improvement of other manifestations of GCA | weeks 4, 8, and 13
  Proportion of patients with improvement of other manifestations of GCA with tocilizumab and prednisone at weeks 4, 8, and 13
biological improvement | weeks 4, 8, and 13
  Proportion of patients with biological improvement (i.e. CRP and ESR) with tocilizumab and prednisone at weeks 4, 8, and 13
recurrence of AION | week 13
  Influence of 1-month tocilizumab treatment on recurrence of AION, at W13.
recurrence of GCA | Week 13
  Influence of 1-month tocilizumab treatment on recurrence of GCA, at Week 13.
first recurrence of GCA | weeks 1, 2, 3, 4, 8 and 13
  Time to first recurrence of GCA
Immunological biomarkers | weeks 0,4 and 13
  Immunological biomarkers of response to Tocilizumab assessed at W0, W4, and W13.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Heron, MD, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vints
Locations (10):
- France (10):
  - CHU de Caen - Hôpital de la Côte de Nacre, Caen
  - Hôpital François Mitterrand, Dijon
  - CHU de Limoges, Limoges
  - CH Montfermeil, Montfermeil
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - Saint-Antoine Hospital, Paris
  - Pitié-Salpetrière Hospital, Paris
  - Cochin Hospital, Paris
  - Fondation Rothschild,, Paris
  - Groupe Hospitalier Diaconesses-Croix Saint Simon,, Paris